CLINICAL TRIAL: NCT04739787
Title: The Relationships of Regular Preoperative Physical Activities Between Postoperative Pain and Postoperative Nausea and Vomiting on Different Type of Surgeries
Brief Title: The Effects of Preoperative Physical Activities on Surgeries
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chiayi Christian Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ChiayiCH
Record Dates: First submitted 2021-01-28; First posted 2021-02-05 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Postoperative Pain; Postoperative Nausea and Vomiting; Prehabilitation; Physical Activities
MeSH Terms: conditions — Pain, Postoperative; Postoperative Nausea and Vomiting; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Recommendation is strong on physical activity (PA) in the prehabilitation of Enhanced Recovery After Surgery (ERAS) for various types of surgeries. The evidence is however weak regarding ERAS protocols. Many studies have showed that physical exercise and PA have hypoalgesic effects on healthy individuals and they have better pain tolerance too. Here the investigators study changes in postoperative pain and postoperative nausea and vomiting for various types of surgical patients after performing preoperative PA at moderate or vigorous intensity Vs non-preoperative PA patients.

DETAILED DESCRIPTION:
Despite the increasing knowledge on the mechanisms of incisional inflammation, transmission of nociception signals, peripheral and central sensitization, and on top of the current advancements in pharmacology, pharmaceutics, techniques and equipment, unfortunately, the US Institute of Medicine revealed that 80% of patients receiving surgery have reported postoperative pain with 88% of them at moderate, severe, or extreme levels. Opioids for postoperative pain are commonly administered to relieve moderate to severe pain, therefore, the postoperative nausea and vomiting (PONV) incidence will be increased.

ERAS is a prevalent policy that combines evidence-based perioperative care to accelerate surgical recovery, Anesthesiologists are involved in many perioperative ERAS elements of patients in terms of evaluation and implementation: e.g., like prehabilitation via education of physical and core muscles training on the pain management clinic, perioperative multi-modal pain management and multi-modal anti-emetic prophylaxis against PONV.

The overarching aim of multimodal structured prehabilitation programs is to increase, for instance, the cardiopulmonary and musculoskeletal preoperative functional reserve, leading to better postoperative functional recovery and a reduced incidence of complications.

Better ischemic pain tolerance is well documented after combined moderate-and vigorous-intensity aerobic exercise for healthy individuals and acute exercise also has hypoalgesic effects.Unfortunately, these physical activity (PA) researchers have not evaluated specifically effects on postoperative pain and PONV.

The goal of our study is to determine the relationship between preoperative PA on postoperative pain and PONV for different types of surgery, that is, breast neoplasms, thoracic, laparoscopic abdominal, abdominal laparotomy, Ears-Nose-Throat, urinary tract stones and tumors, orthopedic, plastic, spinal and colorectal surgeries.

METHODS:

This is a single center, observational retrospective (preoperative PA patients group vs preoperative non-PA patients group) trial. Information on the incidence and severity of pain and PONV of each patient are periodically recorded at time-points of 1, 4, 7, 10 and 24 hours after various types of surgical operation. Our study was aimed to determine beneficial effects on postoperative pain and PONV for patients after performing preoperative PA for 6 to 8 weeks vs non-PA patients. The investigators employed the recommendations of the American College of Sport Medicine and the World Health Organization for adults to divide our PA patients group into moderate-intensity as 30-60 min∙d-1 (≥150 min∙wk-1 ) and vigorous-intensity as 20-60 min∙d-1 (≥75 min∙wk-1). The severity of postoperative pain and PONV were measured at 1, 4, 7, 10 and 24 hours after the surgical operations for the PA patients group and the non-PA patients group. The severity of postoperative pain were recorded by using 0-10 Numeric Rating Scale and postoperative nausea and vomiting after surgeries were measured by using 5 points Likert Scale (1-5) to record the severity of postoperative pain and PONV after different types of surgery.

The operations were performed under general anesthesia (GA) with endotracheal intubation or inhalation through laryngeal mask.

The procedures of GA will be discussed and decided by one of our anesthesiologists of the Chia-Yi Christian Hospital together with patients/caregivers at the Pre-Anesthesia Consultation Clinic. We used the American Society of Anesthesiologists physical status scoring system for risk stratification, the approaches of Apfel's preventive strategy of postoperative nausea and vomiting prophylaxis, perioperative multi-modal pain management in addition to other appropriate elements in ERAS. PONV defined as nausea, vomiting or retching within 24 h of surgery.

The principle investigator is responsible for the data collection of this retrospective study and recorded of the severity of the postoperative pain and PONV at time-points of 1, 4, 7, 10 and 24 hours after various types of surgical operation via the "Postanesthesia Patient Interview and Record Sheet" and the nursing care recorded at the ward for the PA patients group and the non-PA patients group.

ELIGIBILITY:
Inclusion Criteria:

1. aged ≥18 y/o
2. Enrolled in-patients
3. Patients are scheduled to undergo various operations.
4. The surgeries are expected to last ≥60 minutes
5. Endotracheal intubation or laryngeal mask inhalation general anesthesia.

Exclusion Criteria:

1. Patients will transferred to the intensive care unit after operations.
2. American Society of Anesthesiology physical status ≥4
3. poorly controlled diabetic mellitus (HA1c ≥9)
4. prolonged corrected QT interval (male ≥0.45 sec, female ≥0.47 sec)
5. Allergy to any opioids (i.e., morphine, fentanyl, pethidine and others) and nonopioids (i.e., selective or nonselective NSAIDs and acetaminophen)
6. Allergy to dexamethasone, granisetron, droperidol, metoclopramide used for prevention of postoperative nausea and vomiting
7. Deaf or unable to speak/understand Taiwanese or Mandarin
8. Failed to recall or uncertain on how many days/times they had spent doing moderate or vigorous physical activity on recent 6 to 8 weeks before receiving surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population are the preoperative physical activities patients and the preoperative non-physical activities patients.
  One of our registered nurse of our Anesthesiology Department will go to the postoperative patient's ward within 24 hours after their surgeries in order to collect the data of severity of pain, PONV and other discomforts of the patients at time-points of 1, 4, 7, 10 and 24 hours after various types of surgical operation via asking patients/caregivers and the nursing care recorded on the wards for each patient. All of the collected data will be recorded into the "Postanesthesia Patient Interview and Record Sheet" of the Anesthesiology Department.
Sampling Method: Non-Probability Sample
Enrollment: 5500 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The effects of physical activities on postoperative pain | 2 years
  Comparison of the effects of physical activity and non-physical activity patients groups on postoperative pain after different types of surgeries. The severity of postoperative pain is measured by using 0-10 Numeric Rating Scale.
The effects of physical activities on postoperative nausea and vomiting | 2 years
  Comparison of the effects of physical activity and non-physical activity patients groups on postoperative nausea and vomiting (PONV) after different types of surgeries. PONV defined as nausea, vomiting or retching within 24 hours The incidence and severity of PONV are measured by using 5 points Likert Scale (1-5) with 1 represents no any discomfort to 5 represents terribly uncomfortable.